CLINICAL TRIAL: NCT06445855
Title: The Effectiveness of Online Interpersonal Relationships-Based Pyschoeducation in Increasing Sexual Interest and Arousal in Women With Sexual Interest and Arousal Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Zeynep Dilşah Yılmaz, PHD Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Istanbul University-Cerrahpasa
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Sexual Arousal Disorder; Sexual Desire Disorder
Keywords: Sexual Arousal Disorder; Sexual Desire Disorder; Online Intervention Program; Sexual Interest/ Arousal Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Intervention Model Description: One waiting group and one experimental group
Who Masked: Participant, Outcomes Assessor
Masking Description: Women to be included in the study will be divided into two groups after randomization. The first group will be the experimental group and the second group will be the waiting group. The experimental group will receive 8 weeks of interpersonal relationship-based online psychotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Women in the experimental group will receive an 8-week online intervention program based on interpersonal relationships. An internet-based intervention application will be developed for this intervention. All interventions will be implemented from this intervention.
  Interventions: Behavioral: Interpersonal relationship-based intervention program
- Waiting group (Other): After the interventions in the experimental group are completed, the intervention program will be applied to the women in the waiting group.
  Interventions: Behavioral: Interpersonal relationship-based intervention program

INTERVENTIONS:
Behavioral: Interpersonal relationship-based intervention program — An interpersonal relations-based intervention program will be implemented with an online intervention platform.

SUMMARY:
This study will be conducted to examine the effectiveness of interpersonal relationships-based online psychoeducation developed for women with sexual interest and arousal disorders.

DETAILED DESCRIPTION:
Female sexual interest and arousal disorders are common among sexual dysfunctions. In addition to the physical and mental health of women with sexual interest and arousal disorder, interpersonal relationships are also negatively affected. Based on this relationship, it is predicted that interpersonal relationship-based psychoeducation will be effective in the treatment of sexual interest and arousal disorder.

Interpersonal Relationship Psychotherapy or counseling is a short-term, easy, accessible approach that focuses specifically on interpersonal problems and is based on attachment theory, aiming to reduce depressive symptoms and improve interpersonal functioning.

The number of internet users and the possibilities of access to the internet are increasing significantly all over the world, and online health services via the internet are becoming widespread. Online psychoeducation inevitably takes its place in internet-based applications with technological developments.

In this context, this study will be conducted to increase the sexual interest and arousal levels of women with sexual interest and arousal disorders through online psychoeducation.

ELIGIBILITY:
Inclusion Criteria:

* A person of female biological sex,
* Expressing difficulties in sexual interest and arousal (yes to at least three of the following criteria) (questions related to these criteria will be added to the interview form)
* Decrease/absence in frequency or intensity of sexual activity,
* Decrease/absence of sexual fantasies/erotic thoughts,
* Inability to initiate sexual intercourse with their partner,
* Lack of sexual excitement and pleasure in almost all sexual relationships (about 75%),
* Decreased/absence of sexual interest/arousal to internal or external sexual erotic stimuli (e.g. written, oral, visual),
* Decreased/absence of genital or nongenital sensations in almost all sexual relationships (approximately 75%).
* Low mean scores on the Female Sexual Function Index and Sexual Interest and Desire Inventory-Female scales (mean score on the Female Sexual Function Index below 26.55, mean score on the Sexual Interest and Desire Inventory-Female below 33)
* Have sufficient knowledge about the use of the Internet,
* Women who have had a sexual partner for at least 1 year are among the inclusion criteria for this study.

Exclusion Criteria:

* Becoming pregnant or planning pregnancy during the psychoeducation period,
* Receive treatment for any sexual dysfunction,
* Withdrew from the study at any stage of the study,
* Women who do not attend more than one session of the psychoeducation will not be included in the study (Women who miss the weekly program of the psychoeducation will be allowed a maximum of 2 make-up sessions).

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Sexual Interest and Desire Inventory-Female (SIDI-F) | 12 weeks
  The inventory is a 13-item inventory developed to measure the level of sexual interest and arousal of women specifically in the last 4 weeks. A total score between 0 and 51 is obtained from the SIDI-F. The cut-off score of the inventory is 33 and 94.7% of the women below this score have a sexual interest and desire disorder.

SECONDARY OUTCOMES:
Female Sexual Distress Scale-Revised | 12 weeks
  The 13-item scale, which was developed to evaluate the distress experienced by women with sexual dysfunction, has a 5-point Likert structure. The increase in the scale score indicates an increase in the level of sexual distress in women. The cut-off score of the scale is 11.
Female Sexual Function Index (FSFI) | 12 weeks
  The scale was developed to evaluate the sexual problems and sexual functions of individuals in general in the last 4 weeks and consists of 19 questions and 6 subcategories (sexual desire, sexual arousal, lubrication, orgasm, satisfaction and pain). The first 2 questions of the scale are related to "sexual desire", questions 3-6 to "sexual arousal", questions 7-10 to "lubrication", questions 11-13 to "orgasm", questions 14-16 to "satisfaction" and questions 17-19 to "pain" subcategories. Questions 1, 2, 15 and 16 are scored between 1 and 5, while the remaining items are scored between 0 and 5. The highest score that can be obtained from the scale is 36 and the lowest score is 2.
Interpersonal Relationship Dimensions Scale | 12 weeks
  the dimensions of interpersonal relationships. It has four sub-dimensions: dependency, empathy, trust in others and emotional awareness. The higher the score, the higher the related sub-dimension
System Usability Scale (SUS-TR) | 12 weeks
  hardware, mobile devices, online web pages. It is a five-point Likert-type scale with 10 items. Items with odd numbers are scored from one to five, while items with even numbers are scored from five to one. In the scale score calculation, the score obtained from each participant is multiplied by 2.5 and a score between 0-100 is obtained. A high score on the scale indicates that the usability of the system is high.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website address — https://cinselakademi.com/Login